CLINICAL TRIAL: NCT03622138
Title: The Impact Integrated Data System for Quality and Outcomes Tracking of Prevention Programs
Acronym: Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R44MH111299 (NIH)
Record Dates: First submitted 2018-07-10; First posted 2018-08-09 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Trauma, Psychological; Social Skills; Family Dysfunctional
Keywords: Evidence-based Prevention Programs; Youth Prevention Programs; Outcomes Data; Continuous Quality Improvement
MeSH Terms: conditions — Psychological Trauma; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naive EBP Providers (Experimental): Naive Providers (providers with no prior experience implementing the EBP) will attend a one-hour orientation meeting via web-based meeting software (e.g., WebEx) or in person to receive training on research procedures and implementation methods for the study. Participants will complete online surveys via 3C's secure system for any measures not collected directly via Impact. Providers will receive secure login information to the survey system and automatic email alerts with links to surveys to prompt completion. Surveys will be completed at PRE and POST time points to assess feasibility, usability, and value. 3C research staff will be available to assist providers (via email and phone) throughout the pilot field study.
  Interventions: Other: Impact
- Experienced EBP Providers (Experimental): Experienced EBP Providers (providers with prior experience implementing the EBP) will attend a one-hour orientation meeting via web-based meeting software (e.g., WebEx) or in person to receive training on research procedures and implementation methods for the study. Participants will complete online surveys via 3C's secure system for any measures not collected directly via Impact. Providers will receive secure login information to the survey system and automatic email alerts with links to surveys to prompt completion. Surveys will be completed at PRE and POST time points to assess feasibility, usability, and value. 3C research staff will be available to assist providers (via email and phone) throughout the pilot field study.
  Interventions: Other: Impact

INTERVENTIONS:
Other: Impact — Impact is an easy to use, cost- and time-efficient technology platform that is capable of (a) gathering relevant process and outcomes data in a feasible way within real-world service settings; (b) producing real-time analytics (e.g., graphical displays) and meaningful reports at the provider, service setting, and broader levels (e.g., state-wide); and (c) linking data analytics to continuous quality improvement (CQI) feedback to help providers achieve best practices and targeted youth outcomes.

SUMMARY:
There has been substantial progress in developing evidence-based prevention programs (EBPPs) for preventing risky behaviors and promoting positive outcomes for youth. Unfortunately, their adoption, quality implementation, long-term sustainability, and scalability in real world service settings, continues to lag far behind resulting in an inability to achieve the intended broad scale public impact. This SBIR Phase II project will build on the findings and feedback gathered from stakeholders in the Phase I project to fully develop and test the Impact implementation support system. Impact will provide an easy to use, cost- and time-efficient technology platform that is capable of (a) gathering relevant process and outcomes data in a feasible way within real-world service settings; (b) producing real-time analytics (e.g., graphical displays) and meaningful reports at the provider, service setting, and broader levels (e.g., state-wide); and (c) linking data analytics to continuous quality improvement (CQI) feedback to help providers achieve best practices and targeted youth outcomes.

DETAILED DESCRIPTION:
Describe the objective(s) of the proposed research including purpose, research question and design, anticipated length of the entire study, hypothesis and relevant background information.

There has been substantial progress in developing evidence-based prevention programs (EBPPs) for preventing risky behaviors and promoting positive outcomes for youth. Unfortunately, their adoption, quality implementation, long-term sustainability, and scalability in real world service settings, continues to lag far behind resulting in an inability to achieve the intended broad scale public impact. This SBIR Phase II project will build on the findings and feedback gathered from stakeholders in the Phase I project to fully develop and test the Impact implementation support system. Impact will provide an easy to use, cost- and time-efficient technology platform that is capable of (a) gathering relevant process and outcomes data in a feasible way within real-world service settings; (b) producing real-time analytics (e.g., graphical displays) and meaningful reports at the provider, service setting, and broader levels (e.g., state-wide); and (c) linking data analytics to continuous quality improvement (CQI) feedback to help providers achieve best practices and targeted youth outcomes.

For this Phase II project, 3C will create three instantiations (or 'instances') of Impact, i.e., one instance for each of three EBPPs. These EBPPs explicitly target one or more mental health outcomes for youth, and provide a test of the application of Impact to a variety of service delivery models, including small group-based, universal classroom, and parent training:

1. Cognitive Behavioral Intervention for Trauma in Schools (CBITS) is an evidence-based program delivered by mental health providers in the school setting. CBITS has been shown to reduce posttraumatic stress disorder (PTSD) symptoms, depression, and anxiety for youth in grades 5-12 as well as improve psychosocial functioning. The 10-session program teaches cognitive behavioral skills using a mixture of didactic presentations, relaxation training, and strategies to combat negative thoughts, reduce avoidance, develop a trauma narrative, and build social problem solving skills. CBITS also includes 1-3 individual child sessions and 2 optional parent sessions.
2. Social Skills Group Intervention K-2 (S.S. GRIN K-2) is an evidence-based program delivered by mental health providers in the school setting to kindergarten through 2nd grade children. S.S. GRIN has been shown to improve self-esteem and self-efficacy, as well as reduce social anxiety and, in aggressive children, reduce aggression and bullying behavior. The intervention includes 10 small group sessions, delivered in an in-person format.
3. The third EBP that will be developed and tested for this Phase II research is Strengthening Families, which has been shown to improve youth outcomes related to substance use, aggressive and hostile behaviors, and risky sexual behaviors, as well as parent protective factors such as affective quality and general child management. The program includes 10-14 sessions, each of which consists of a separate parent and child meeting followed by a family meeting, designed to help families improve communication, conflict resolution, appropriate disciplinary factors, and child involvement in the family. Strengthening Families is implemented in schools, community centers, and mental health facilities by two to four mental health providers.

The proposed three-year project will accomplish three specific aims: (1) fully develop the Impact software platform for the three Blueprints-supported EBPPs listed above, (2) conduct a pilot field study to test whether and in what ways Impact is superior to currently used process and outcomes tracking methods for each EBPP, and (3) prepare Impact for commercialization.

Impact's technology infrastructure will be able to accommodate a wide array of EBPPs, providing a much needed cost-effective mechanism to support broad-scale dissemination and use in service settings. In addition, administrators will be able to track implementation, thus enhancing accountability and providing on-going quality assurance, while also providing data analytics to quickly and effectively monitor impact and cost-effectiveness, thereby increasing the likelihood a program's core features are adhered to over time and maximizing treatment benefits for youth.

ELIGIBILITY:
Inclusion Criteria:

* Must be an Evidence-based Prevention Program Provider
* Regularly implement one of the three supported EBPPs to youth in a school or community setting
* Commit to implementing that EBPP over the study period (approximately one school year)
* Serve a minimum of 10 youth over the study period
* Be willing to allow 3C researchers to collect data from their setting

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Fidelity to the Program Model | To assess change, this measure will be taken each time providers enter data into the Impact system after each session (once per week for up to 12 weeks).
  Providers will complete a Fidelity form, and will receive a total score ranging from 0 to 100, with 80 or higher representing better outcomes. Scores are calculated by converting responses (1 to 5) to percentage (0 to 100) and averaging item percentages.

SECONDARY OUTCOMES:
Attitudes toward EBP Tracking | To assess change, this measure will be taken (1) at baseline (PRE) and (2) following completion of providers' use of Impact, up to 9 months (POST).
  Providers will complete the 22-item Attitudes Towards Standardized Assessment scale which measures provider perceptions of using data in practice. Three subscale scores will be calculated by averaging responses of each item within that subscale. Scores range from 1=Strongly Agree to 5=Strongly Disagree with 5 being the better outcome.
Skilled Use of Data | To assess change, this measure will be taken (1) at baseline (PRE) and (2) following completion of providers' use of Impact, up to 9 months (POST).
  Providers will rate their understanding of and skill using data for an EBP using an 8-item Skilled Use of Data scale, measuring self-reported skill level for using data related to an EBP. Scores range from 1=Minimal to 5=Advanced, with 5 being the better outcome. A total score is calculated by averaging responses for each item.
Satisfaction with Impact assessed by Acceptability Scale | This evaluation measure will be assessed following completion of providers' use of Impact, up to 9 months (POST).
  Providers will rate their satisfaction with using Impact as a method to enter and track data using an 80-item Acceptability scale across 10 domains. A subscale score will be calculated for each domain by averaging scores for each item within that domain. Scores range from 1=Definitely No to 5=Definitely Yes, with 5 being the better outcome.
Practicality of Impact | This evaluation measure will be assessed following completion of providers' use of Impact, up to 9 months (POST).
  Providers will complete a Practicality evaluation scale (80 items across 10 domains). A score will be calculated for each domain, for a total of 10 subscale scores. Each subscale score ranges from 1=Very Low to 7=Very High, with 7 being the better outcome. Subscale scores are calculated by averaging the item responses within each subscale.
Integration of Impact | This evaluation measure will be assessed following completion of providers' use of Impact, up to 9 months (POST).
  Providers will complete an 8-item evaluation scale (Integration of Impact) measuring how well Impact works with other systems. A total score for this scale will be calculated by averaging item responses, and scores range from 1=Strongly Disagree to 7=Strongly Agree, where 7 is the better outcome.
Usability of Impact | This evaluation measure will be assessed following completion of providers' use of Impact, up to 9 months (POST).
  Providers will complete a 20-item Usability scale adapted from the Post-Study System Usability Questionnaire (PSSUQ). Three subscale scores will be calculated, and each ranges from 7=Strongly Disagree to 1=Strongly Agree, with 1 being the better outcome. Scores are calculated by averaging item responses within each subscale.
Value of Impact | This evaluation measure will be assessed following completion of providers' use of Impact, up to 9 months (POST).
  Providers will complete the 8-item Value of Impact scale, and a total score will be calculated by averaging item responses. Scores range from 1=Poor to 5=Excellent, with 5 being the better outcome.
Commitment to Change | This evaluation measure will be assessed following completion of providers' use of Impact, up to 9 months (POST).
  Providers will complete the 18-item Commitment to Change scale, which measures how committed providers are to use Impact in their organization. Three subscale scores are calculated, and each score ranges from 1=Strongly Disagree to 7=Strongly Agree, with 7 being the better outcome. Scores are calculated by averaging item responses within each subscale.
Time Spent Using Impact | This measure will be assessed each week while providers are implementing the EBP and using the Impact system (once per week, up to 12 weeks).
  Providers will report the amount of time it takes them to complete all activities (e.g., data entry, generating reports) using Impact. Time will be reported in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa E DeRosier, PhD, Principal Investigator — 3C Institute
Locations (1):
- 3C Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided